CLINICAL TRIAL: NCT04335747
Title: COVID-19 Infection in Vulnerable Patients With Inflammatory Rheumatic Diseases
Status: Terminated | Type: Observational
Why Stopped: Low recruitment rate
Sponsor: Salome Kristensen (Other)
Responsible Party: Sponsor-Investigator, Salome Kristensen, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: 20200401
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis; Systemic Lupus Erythematosus; Giant Cell Arteritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis; Lupus Erythematosus, Systemic; Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients with inflammatory rheumatic diseases who are hospitalised due to a COVID-19 infection
  Interventions: Other: COVID-19 infection
- Group 2: Patients without inflammatory diseases who are hospitalised due to a COVID-19 infection
  Interventions: Other: COVID-19 infection
- Group 3: Patients with inflammatory rheumatic diseases who are having routine blood samples taken under the COVID-19 epidemic after inclusion and who have NOT been hospitalised due to a COVID-19 infection
- Group 4: Healthy subjects from the Danish Blood Donors have NOT been hospitalised due to a COVID-19 infection

INTERVENTIONS:
Other: COVID-19 infection — Hospitalisation due to a confirmed COVID-19 infection
  Groups: Group 1; Group 2

SUMMARY:
The trial is a prospective, observational study aiming to identify risk factors for serious COVID-19 infection by evaluating clinical measures and biomarkers of inflammation in patients with inflammatory rheumatic disease hospitalized with COVID-19 compared with control groups.

DETAILED DESCRIPTION:
The pandemic caused by the coronavirus, SARS-CoV-19, has severely affected health care systems around the world. In Denmark, more than 85,000 patients have a diagnosis of rheumatoid arthritis (RA), psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus (SLE), or giant cell arthritis, and many are treated with immunosuppressive therapy including biologics.

At present it is unclear whether the best course of action during a viral pandemic is to pause treatment with biologics, change to drugs with a different mode of action or continue treatment as usual.

Many patients with RA and SLE receive hydroxychloroquine (HCL) treatment for their rheumatic disease, but HCL has also been suggested as a potential treatment for COVID-19 infection.

This trial aim to identify risk factors for serious COVID-19 infection by evaluating clinical measures and biomarkers of inflammation, including IL6 and IL10 in patients with inflammatory rheumatic disease hospitalized with COVID-19 compared with measures in control groups.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Diagnosed with RA, PsA, axSpA, SLE or AT and currently treated with either conventional synthetic disease modifying antirheumatic drugs (csDMARDs), biologic disease modifying antirheumatic drugs (bDMARDs), targeted synthetic disease modifying antirheumatic drugs (tsDMARDs) or prednisolone.
* Diagnosed with COVID-19 verified by Polymerase Chain Reaction (PCR) or other accepted methods and hospitalized.
* NOT diagnosed with disease known to cause either immunodeficiency or modification (Human Immunodeficiency Virus [HIV], lymphoproliferative disease etc.).
* Patients (≥18 years).
* Ability and willingness to give written informed consent.
* Ability to cooperate with research staff.

Group 2:

* NOT diagnosed with an inflammatory disease
* NOT treated with either csDMARDs, bDMARDs, tsDMARDs during the past 6 months or current oral prednisolone treatment.
* Diagnosed with COVID-19 verified by PCR or other accepted methods and hospitalized.
* NOT diagnosed with disease known to cause either immunodeficiency or modification (HIV, lymphoproliferative disease etc.).
* Patients (≥18 years).
* Ability and willingness to give written informed consent.
* Ability to cooperate with research staff.

Group 3:

* Diagnosed with RA, PsA, axSpA, SLE or AT and currently treated with either csDMARDs, bDMARDs, tsDMARDs or prednisolone.
* NOT hospitalised due to a COVID-19 infection.
* NOT diagnosed with disease known to cause either immunodeficiency or modification (HIV, lymphoproliferative disease etc.).
* Patients (≥18 years).
* Ability and willingness to give written informed consent.
* Ability to cooperate with research staff.

Group 4:

* Healthy subjects from the Danish Blood Donors.
* Patients (≥18 years).
* NOT diagnosed with an inflammatory disease.
* NOT treated with either csDMARDs, bDMARDs, tsDMARDs during the past 6 months or current oral prednisolone treatment.
* NOT hospitalised due to a COVID-19 infection.
* Ability and willingness to give written informed consent.
* Ability to cooperate with research staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups 1 and 2: admitted patients with a COVID-19 infection at Aalborg University Hospital Group 3: the Rheumatology Outpatient Clinic at Aalborg University Hospital Group 4: the Blood Bank for Danish Blood Donors at Aalborg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Disease activity | Last registration of disease activity in the medical journal before admission/inclusion
  The objective is to examine whether increased disease activity leads to increased risk of hospitalization due to COVID-19 in patients with inflammatory rheumatic disease

SECONDARY OUTCOMES:
Immune modulating treatments | Current immune modulating treatments at admission/inclusion
  Examine whether immune modulating treatments protect or leads to increased risk of hospitalization due to COVID-19 in patients with inflammatory rheumatic disease.
Biomarkers | Blood sample 1 is taken 0-3 days after inclusion and blood sample 2 is taken 2-6 weeks after blood sample 1
  Identify prognostic biomarkers by comparing serology of patients with inflammatory rheumatic disease hospitalized with COVID-19 and comparing them with the two control groups

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, PhD, Principal Investigator — Department of Rheumatology, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No